CLINICAL TRIAL: NCT04783688
Title: Evaluation of a Full Face Snorkel Mask (FFSM)
Brief Title: Evaluation of Full Face Snorkel Masks (FFSMs)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Divers Alert Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00106241
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-03

CONDITIONS: Snorkeling; Face Mask Squeeze; Underwater Physiology; Swimming Physiology

STUDY DESIGN:
Intervention Model Description: Study is a measurement of subjects performing normal tasks in a controlled environment, with physiological measurements
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): All subjects will snorkel using the same FFSMs.
  Interventions: Other: Full Face Snorkel Mask (FFSM)

INTERVENTIONS:
Other: Full Face Snorkel Mask (FFSM) — A mask used for snorkeling that covers the entire face, as opposed to a conventional snorkel, which is held in the mouth only.

SUMMARY:
Recently, multiple models of Full Face Snorkel Mask (FFSM) have entered the retail market. However, several fatalities have been reported to the non-profit agency Divers Alert Network (DAN) for snorkelers who were using FFSMs, and most of these fatality reports have unclear or unreported causes of death. This project is to determine the characteristics of the FFSMs when they are in use by snorkelers. Volunteers will be asked to snorkel in a water tank while breathing through several models of commercially available FFSM, one at at time.

DETAILED DESCRIPTION:
The scientific testing will take place in the water tank of Foxtrot chamber at the Duke Center for Hyperbaric Medicine & Environmental Physiology. This Center (referred to as "Duke Hyperbarics") has a long history of testing various aspects of undersea physiology and causes of injury and death. Duke Hyperbarics will conduct the physical tests, and DAN (Divers Alert Network) personnel will also supervise the scientific testing.

The experimental test subjects will be divided into two categories. Before testing, both categories will come in for a screening day, where they will go through the informed consent process and be medically screened for safety to perform activity. For the first category of subjects (Group A), five volunteer subjects will be recruited with no restrictions on age or fitness level. An effort will be made to include representative test subjects from older age ranges (>35 years old) in this group. To ensure they can safely perform light activity, they will be screened for cardiovascular disease, both by questionnaire and by a physical exam during the screening day.

The second group (Group B) will be age 18-40, non-smoking, and screened for fitness using a physical exam and a VO2max test. The reason for these two groups is to ensure that a spectrum of test subjects is examined across the comprehensive range of ages and fitness levels that may participate in snorkeling as recreation.

The testing will be designed to assess the function of the FFSMs produced by multiple brands compared to each other as well as compared to conventional snorkels. Test subjects will be positioned horizontally in warm water. They will be face-down on a bicycle ergometer, grasping handlebars for stability. On the test day, each subject will undergo three test procedures, using first a conventional snorkel then two different brands of FFSM while pedaling the underwater bicycle. Group A will be asked to pedal at a rate that is comfortable for them, while Group B will be given a targeted higher work rate to achieve.

For each FFSM test, the test subject will be asked to place the mask on themselves but provided no further instruction. The pressure exerted by the mask on the forehead will also be measured by placing a small, flexible, force-sensitive gauge between the skirt and the skin (this gauge needs to be in place for only a few seconds and will be removed before snorkeling). At the end of each test, the subjects will be asked to remove the FFSM quickly in response to an audible or visual alarm that will appear three times at randomized intervals. Their ability to remove the masks quickly will be timed.

ELIGIBILITY:
GROUP A:

Inclusion Criteria:

* Preferred >35 years old
* Safe to perform light activity

Exclusion Criteria:

* Subjects must NOT be certified SCUBA divers

GROUP B:

Inclusion Criteria:

* Age 18-40
* VO2max exercise test results >30 mL/kg/min for female, >35 mL/kg/min for male

Exclusion Criteria:

* Subjects must NOT be certified SCUBA divers
* May not be active smokers

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-06-11 (Actual)

PRIMARY OUTCOMES:
Fractional level of oxygen in the breathing gas (at steady state) provided by the different mask models | Estimated 4 hours long
  The breathing gas provided to the snorkeler by the masks will be measured continuously throughout the experiment using a mass spectrometer.
Fractional level of carbon dioxide in the breathing gas (at steady state) provided by the different mask models | Estimated 4 hours long
  The breathing gas provided to the snorkeler by the masks will be measured continuously throughout the experiment using a mass spectrometer.

SECONDARY OUTCOMES:
Speed of removal of the different FFSM models | Estimated 20 minutes
  The speed at which subjects can remove the different models of FFSM will be timed and measured in seconds for comparison between models.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Lance, PhD, Principal Investigator — Duke University Health System, Department of Anesthesiology
Locations (1):
- Duke University Center for Hyperbaric Medicine & Environmental Physiology, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Processed, anonymized experimental results will be shared with Divers Alert Network (DAN).